CLINICAL TRIAL: NCT06252285
Title: Phase III, Randomized, Observer-blind, Placebo-controlled, Multi-center, Multinational Study to Evaluate the Efficacy, Immunogenicity, and Safety of a Respiratory Syncytial Virus Vaccine in Infants and Toddlers (PEARL)
Brief Title: Efficacy, Immunogenicity, and Safety Study of a Respiratory Syncytial Virus Vaccine in Infants and Toddlers
Acronym: PEARL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAD00004; 2023-505762-29 (Registry Identifier: CTIS); U1111-1280-7192 (Registry Identifier: ICTRP); VAD00004 (Other: Sanofi Identifier)
Record Dates: First submitted 2024-01-24; First posted 2024-02-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: RSV Immunisation
MeSH Terms: interventions — YM 534

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * Blinding for vaccine group assignment: participants, parents or legally acceptable representatives (LARs), outcome assessors, investigators, laboratory personnel, Sponsor study staff
  * No blinding for study staff who prepare and administer the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 RSVt Vaccine (Experimental): Participants will receive 2 intranasal administrations of RSVt vaccine
  Interventions: Biological: RSVt Vaccine
- Group 2 Control (Placebo Comparator): Participants will receive 2 intranasal administrations of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSVt Vaccine — Pharmaceutical form:Suspension of virus in a nasal spray-Route of administration:Intranasal
  Other Names: 534
  Arms: Group 1 RSVt Vaccine
Biological: Placebo — Pharmaceutical form:Suspension of virus in a nasal spray-Route of administration:Intranasal
  Arms: Group 2 Control

SUMMARY:
This study is a phase III, randomized, observer-blind, placebo-controlled, multinational, multi-center study to be conducted in approximately 6300 children 6 months to < 22 months of age. The purpose of the study is to evaluate the efficacy, immunogenicity, and safety of Respiratory Syncytial Virus Toddler (RSVt) vaccine administered by intranasal route compared to placebo.

Eligible participants will be randomized in a 1:1 ratio to receive 2 intranasal administrations of either the RSVt vaccine or placebo.

Study duration will be 24 months for each participant. The safety follow-up will start after the first vaccination and up to the end of the study.

DETAILED DESCRIPTION:
Study duration will be 24 months for each participant. The safety follow-up will start at inclusion and up to the end of the study.

ELIGIBILITY:
Inclusion Criteria: -Aged 6 months to < 22 months on the day of inclusion (means the day of the 6-month birthday to the day before the 22-month birthday)

* Participants who are healthy as determined by medical evaluation including medical history
* Born at full term of pregnancy (≥ 37 weeks)

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* History of medically diagnosed wheezing
* Any acute febrile illness in the past 48 hours that according to investigator judgment is significant enough to interfere with successful inoculation on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Probable or confirmed ongoing case of viral respiratory infection (including COVID-19, influenza, rhinovirus, etc.) at the time of enrollment. A prospective participant should not be included in the study until the respiratory infection has resolved.
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is HIV infected
  * a person who has received chemotherapy within the 12 months prior to study enrollment
  * a person who has received (within the past 6 months) or is receiving (at the time of enrollment) immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Potential close contact with other immunocompromised individual within 30 days after each vaccination as per investigator's discretion
* Participant's biological mother's previous receipt or planned administration of an investigational RSV vaccine during pregnancy and/or breastfeeding.
* Receipt or planned receipt of any of the following vaccines prior to enrollment or after the first study intervention administration:

  * Any other intranasal live attenuated vaccine within the 28 days prior to and after Dose 1 study administration
  * Unless given on the day of Dose 1 study administration, any other injectable live attenuated vaccines within the 28 days prior to and after. Concomitant receipt on the day of Dose 1 study administration is allowed.
* Previous receipt of an investigational RSV vaccine or receiving any anti-RSV product (such as ribavirin or RSV immune globulin) at the time of enrollment. Previous receipt of an RSV monoclonal antibody within 6 months prior to the first study vaccine administration.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of intranasal and intra-ocular medications within 3 days prior to study enrollment
* Participation at the time of study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6300 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of lower respiratory tract disease (LRTD) (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of LRTD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)

SECONDARY OUTCOMES:
Occurrence of upper respiratory tract disease (URTD) (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of URTD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of LRTD (during RSV Season 1) associated with any RT PCR confirmed RSV strain leading to hospitalization > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of LRTD associated with any RT PCR confirmed RSV strain leading to hospitalization, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of severe LRTD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of severe LRTD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of urgent care visits, associated with an episode of LRTD over RSV Season 1, associated with any RT-PCR confirmed RSV strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of urgent care visit associated with an episode of LRTD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of acute respiratory disease (ARD) (during RSV Season 1) associated with any RT-PCR confirmed RSV strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of ARD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of hospitalizations, associated with an episode of ARD over RSV Season 1, associated with any RT-PCR confirmed RSV strain > 21 days post dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of hospitalizations associated with an episode of ARD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of urgent care visits, associated with an episode of ARD over RSV Season 1, associated with any RT-PCR confirmed RSV strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of urgent care visit associated with an episode of ARD associated with any RT PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1
Occurrence of LRTD (during RSV Season 1) associated with an RT-PCR confirmed RSV A or B strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of LRTD associated with an RT PCR confirmed RSV A or B, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of URTD (during RSV Season 1) associated with an RT-PCR confirmed RSV A or B strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of URTD associated with an RT-PCR confirmed RSV A or B, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of ARD (during RSV Season 1) associated with an RT PCR confirmed RSV A or B strain > 21 days post-dose 2 | from 22 days post-dose 2 up to the start date of first occurrence of ARD associated with an RT-PCR confirmed RSV A or B, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of LRTD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 1 | from 22 days post-dose 1 up to the start date of first occurrence of LRTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of URTD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 1 | from 22 days post-dose 1 up to the start date of first occurrence of URTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of ARD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 1 | from 22 days post-dose 1 up to the start date of first occurrence of ARD associated with any RT-PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of LRTD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 2, in RSV-exposed participants | from 22 days post-dose 2 up to the start date of first occurrence of LRTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1
Occurrence of URTD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 2, by baseline serostatus | from 22 days post-dose 2 up to the start date of first occurrence of URTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of ARD (during RSV Season 1) associated with any RT PCR confirmed RSV strain > 21 days post-dose 2, by baseline serostatus | from 22 days post-dose 2 up to the start date of first occurrence of ARD associated with any RT-PCR confirmed RSV strain, assessed up to the end of RSV season 1 (ie. up to 12 months post-dose 1)
Occurrence of LRTD (during RSV Season 2), associated with any RT-PCR confirmed RSV strain | from 12 months post-dose 1 up to the start date of first occurrence of LRTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of the study (ie. up to 24 months post-dose 1)
Occurrence of URTD (during RSV Season 2), associated with any RT-PCR confirmed RSV strain | from 12 months post-dose 1 up to the start date of first occurrence of URTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of the study (ie. up to 24 months post-dose 1)
Occurrence of ARD (during RSV Season 2), associated with any RT PCR confirmed RSV strain | from 12 months post-dose 1 up to the start date of first occurrence of ARD associated with any RT-PCR confirmed RSV strain, assessed up to the end of the study (ie. up to 24 months post-dose 1
Occurrence of LRTD (during RSV Season 2), associated with any RT PCR confirmed RSV strain, by baseline serostatus | from 12 months post-dose 1 up to the start date of first occurrence of LRTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of the study (ie. up to 24 months post-dose 1)
Occurrence of URTD (during RSV Season 2), associated with any RT PCR confirmed RSV strain, by baseline serostatus | from 12 months post-dose 1 up to the start date of first occurrence of URTD associated with any RT-PCR confirmed RSV strain, assessed up to the end of the study (ie. up to 24 months post-dose 1)
Occurrence of ARD (during RSV Season 2), associated with any RT PCR confirmed RSV strain, by baseline serostatus | from 12 months post-dose 1 up to the start date of first occurrence of ARD associated with any RT-PCR confirmed RSV strain, assessed up to the end of the study (ie. up to 24 months post-dose 1)
Presence of solicited administration site reactions within 21 days after each vaccination | Within 21 days after each vaccination
  Number of participants experiencing solicited site reactions
Presence of solicited systemic reactions within 21 days after each vaccination | Within 21 days after each vaccination
  Number of participants experiencing solicited systemic reactions
Presence of unsolicited systemic adverse events (AEs) reported in the 30 minutes after each vaccination | Within 30 minutes after each vaccination
  Number of participants experiencing immediate unsolicited systemic AES
Presence of unsolicited AEs within 28 days after each vaccination | Within 28 days after each vaccination
  Number of participants experiencing unsolicited AES
Presence of medically attended adverse events MAAEs throughout the study | Throughout the study (approximately 24 months)
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) throughout the study | Throughout the study (approximately 24 months)
  Number of participants experiencing SAEs
Presence of adverse events of special interest (AESIs) throughout the study | Throughout the study (approximately 24 months)
  Number of participants experiencing AESIs
RSV A serum neutralizing antibody titers at D01 | Day 01
  Antibody titers are expressed as GMTs at baseline
RSV B serum neutralizing antibody titers at D01 | Day 01
  Antibody titers are expressed as GMTs at baseline
RSV A serum neutralizing antibody titers at 28 days post-dose 2 | 28 days post-dose 2
  Antibody titers are expressed as GMTs at post-baseline
RSV B serum neutralizing antibody titers at 28 days post-dose 2 | 28 days post-dose 2
  Antibody titers are expressed as GMTs post-baseline
RSV serum anti-F Immunoglobulin A (IgA) Electrochemiluminescence (ECL) antibody titers at D01 | Day 01
  Antibody titers are expressed as GMTs at baseline
RSV serum anti-F IgG ECL antibody titers at D01 | Day 01
  Antibody titers are expressed as GMTs at baseline
RSV serum anti-F Immunoglobulin A (IgA) ECL antibody titers at 28 days post-dose 2 | 28 Days post-dose 2
  Antibody titers are expressed as GMTs post-baseline
RSV serum anti-F IgG ECL antibody titers at 28 days post-dose 2 | 28 Days post-dose 2
  Antibody titers are expressed as GMTs post-baseline

CONTACTS AND LOCATIONS:
Locations (130):
- United States (50):
  - Central Research Associates - Flourish - PPDS- Site Number : 8400009, Birmingham, Alabama
  - Lakeview Clinical Research- Site Number : 8400024, Guntersville, Alabama
  - Novak Clinical Research- Site Number : 8400069, Tucson, Arizona
  - Madera Family Medical Group- Site Number : 8400029, Madera, California
  - Integrated Clinical Research- Site Number : 8400056, Tarzana, California
  - National Institute of Clinical Research - Victorville - Hesperia Road- Site Number : 8400040, Victorville, California
  - Moore Clinical Research - Brandon- Site Number : 8400065, Brandon, Florida
  - Invictus Clinical Research Group- Site Number : 8400035, Coconut Creek, Florida
  - Site Number : 8400031, Doral, Florida
  - Nona Pediatric Center- Site Number : 8400068, Orlando, Florida
  - Teena Hughes Pediatrics- Site Number : 8400042, Tampa, Florida
  - Morehouse School of Medicine - Atlanta- Site Number : 8400037, Atlanta, Georgia
  - Emory-Children's Center- Site Number : 8400001, Atlanta, Georgia
  - Agile Clinical Research Trials- Site Number : 8400015, Atlanta, Georgia
  - Tekton Research, LLC - 4961 Buford Hwy - Georgia - PPDS- Site Number : 8400064, Chamblee, Georgia
  - Velocity Clinical Research - (Macon - Georgia) - PPDS- Site Number : 8400041, Macon, Georgia
  - iResearch Savannah - CenExel - PPDS- Site Number : 8400032, Savannah, Georgia
  - Medical Research Partners - Ammon- Site Number : 8400059, Ammon, Idaho
  - Clinical Research Prime- Site Number : 8400013, Idaho Falls, Idaho
  - Leavitt Women's Healthcare- Site Number : 8400033, Idaho Falls, Idaho
  - Snake River Research- Site Number : 8400046, Idaho Falls, Idaho
  - Michigan Institute of Research- Site Number : 8400055, Allen Park, Michigan
  - Vida Clinical Studies - Dearborn Heights- Site Number : 8400072, Dearborn Heights, Michigan
  - Great Lakes Research Institute- Site Number : 8400060, Southfield, Michigan
  - Clinical Research Institute - Minneapolis- Site Number : 8400011, Minneapolis, Minnesota
  - Boeson Research - Great Falls- Site Number : 8400008, Great Falls, Montana
  - Velocity Clinical Research - Grand Island- Site Number : 8400017, Grand Island, Nebraska
  - Be Well Clinical Studies - Lincoln- Site Number : 8400058, Lincoln, Nebraska
  - Velocity Clinical Research (Norfolk - Nebraska) - PPDS- Site Number : 8400038, Norfolk, Nebraska
  - Quality Clinical Research - Omaha - Regency Circle- Site Number : 8400016, Omaha, Nebraska
  - Velocity Clinical Research - Omaha- Site Number : 8400054, Omaha, Nebraska
  - Prime Global Research, Inc.- Site Number : 8400043, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400063, Cincinnati, Ohio
  - Senders Pediatrics- Site Number : 8400006, South Euclid, Ohio
  - Cyn3rgy Research- Site Number : 8400014, Gresham, Oregon
  - Medical University of South Carolina - Charleston - Jonathan Lucas Street- Site Number : 8400036, Charleston, South Carolina
  - Palmetto Pediatrics- Site Number : 8400012, North Charleston, South Carolina
  - Parkside Pediatrics - Simpsonville- Site Number : 8400071, Simpsonville, South Carolina
  - Clinical Research Associates Inc- Site Number : 8400005, Nashville, Tennessee
  - Tekton Research, LLC - Beaumont - PPDS- Site Number : 8400061, Beaumont, Texas
  - South Texas Urgent Care - Del Rio- Site Number : 8400062, Del Rio, Texas
  - Ventavia Research Group - Fort Worth- Site Number : 8400022, Fort Worth, Texas
  - Private Practice - Dr. Chinyere N. Awa- Site Number : 8400066, Houston, Texas
  - DM Clinical Research - CyFair Clinical Research Center- Site Number : 8400044, Houston, Texas
  - Maximos Ob/Gyn- Site Number : 8400023, League City, Texas
  - Pediatric Center - Richmond- Site Number : 8400019, Richmond, Texas
  - Tekton Research - FM78- Site Number : 8400067, San Antonio, Texas
  - Alliance for Multispecialty Research - Layton - North Robins Drive- Site Number : 8400030, Layton, Utah
  - Wee Care Pediatrics - Roy- Site Number : 8400002, Roy, Utah
  - Wee Care Pediatrics - Syracuse- Site Number : 8400004, Syracuse, Utah
- Argentina (7):
  - Investigational Site Number : 0320007, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320003, Río Cuarto, Córdoba Province
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320004, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320002, SAN Miguel de Tucumã¡n, Tucumán Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires
- Brazil (8):
  - Obras Sociais Irmã Dulce - Patamares- Site Number : 0760009, Salvador, Estado de Bahia
  - Freire Pesquisa Clínica - Belo Horizonte - Rua Piauí- Site Number : 0760001, Belo Horizonte, Minas Gerais
  - Hospital de Clinicas de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles- Site Number : 0760007, Porto Alegre, Rio Grande do Sul
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP - PPDS- Site Number : 0760010, Ribeirão Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto- Site Number : 0760006, São José do Rio Preto, São Paulo
  - Escola Paulista De Medicina- Site Number : 0760002, Vila Clementino, São Paulo
  - Centro Paulista de Investigaçăo Clínica - CEPIC- Site Number : 0760004, São Paulo
- Chile (3):
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Port Montt
- Investigational Site Number : 1560009, Jiangsu, China
- Colombia (3):
  - Investigational Site Number : 1700004, Acacías
  - Investigational Site Number : 1700002, Chía
  - Investigational Site Number : 1700003, Girardot
- Finland (8):
  - Investigational Site Number : 2460003, Espoo
  - Investigational Site Number : 2460005, Helsinki
  - Investigational Site Number : 2460008, Jarvenpaa
  - Investigational Site Number : 2460004, Kokkola
  - Investigational Site Number : 2460002, Oulu
  - Investigational Site Number : 2460006, Seinäjoki
  - Investigational Site Number : 2460009, Tampere
  - Investigational Site Number : 2460001, Turku
- Japan (11):
  - Investigational Site Number : 3920008, Lizuka-shi, Fukuoka
  - Investigational Site Number : 3920011, Sapporo, Hokkaido
  - Investigational Site Number : 3920007, Kawagoe, Saitama
  - Investigational Site Number : 3920010, Shizuoka-Shi Aoi-Ku, Shizuoka
  - Investigational Site Number : 3920006, Edogawa-Ku, Tokyo
  - Investigational Site Number : 3920001, Fukui
  - Investigational Site Number : 3920002, Fukui-shi
  - Investigational Site Number : 3920004, Fukuoka
  - Investigational Site Number : 3920003, Kagoshima
  - Investigational Site Number : 3920005, Kasuga-Shi
  - Investigational Site Number : 3920009, Osaka
- Kenya (5):
  - Investigational Site Number : 4040007, Butere
  - Investigational Site Number : 4040002, Kisumu
  - Investigational Site Number : 4040003, Kisumu
  - Investigational Site Number : 4040001, Nairobi
  - Investigational Site Number : 4040006, Nairobi
- Mexico (3):
  - Investigational Site Number : 4840008, Monterrey, Nuevo León
  - Investigational Site Number : 4840007, Mexico City
  - Investigational Site Number : 4840004, Veracruz
- Nepal (3):
  - Investigational Site Number : 5240003, Dhulikhel N.p, Bagmati
  - Investigational Site Number : 5240001, Kathmandu, Bagmati
  - Investigational Site Number : 5240002, Nepalgunj, Bheri
- Puerto Rico (4):
  - Clinical Research Investigator Group- Site Number : 6300001, Bayamón
  - Clinical Research Puerto Rico (CRPR), Inc. - Guayama- Site Number : 6300005, Guayama
  - Caribbean Medical Research Center- Site Number : 6300003, San Juan
  - Hospital Pediatrico Universitario- Site Number : 6300002, San Juan
- South Africa (9):
  - Investigational Site Number : 7100007, Brits
  - Investigational Site Number : 7100008, City of Cape Town
  - Investigational Site Number : 7100001, East London
  - Investigational Site Number : 7100005, Johannesburg
  - Investigational Site Number : 7100004, Johannesburg
  - Investigational Site Number : 7100003, Johannesburg
  - Investigational Site Number : 7100006, Paarl
  - Investigational Site Number : 7100002, Pretoria
  - Investigational Site Number : 7100009, Soshanguve
- Spain (5):
  - Investigational Site Number : 7240004, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240001, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240003, Móstoles, Madrid
  - Investigational Site Number : 7240005, Pamplona, Navarre
  - Investigational Site Number : 7240002, Seville, Sevilla
- Thailand (6):
  - Investigational Site Number : 7640002, Bangkok
  - Investigational Site Number : 7640005, Bangkok
  - Investigational Site Number : 7640004, Bangkok
  - Investigational Site Number : 7640001, Chiang Mai
  - Investigational Site Number : 7640006, Hat Yai
  - Investigational Site Number : 7640003, Khon Kaen
- United Kingdom (4):
  - Investigational Site Number : 8260003, Hayle, Cornwall
  - Investigational Site Number : 8260005, Exeter, Devon
  - Investigational Site Number : 8260007, Southampton, Hampshire
  - Investigational Site Number : 8260004, Bristol

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAD00004 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25613&tenant=MT_SNY_9011